CLINICAL TRIAL: NCT03995862
Title: Evaluation of Pre-Exposure Prophylaxis Against HIV in Alpine Region
Acronym: PrEP2A
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Other Study IDs: 18-39-PrEP2A; 2018-A02993-52 (Other: ANSM)
Record Dates: First submitted 2019-06-14; First posted 2019-06-24 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Pre-Exposure Prophylaxis; HIV Seronegativity; Drug Combination
Keywords: tenofovir disoproxil fumarate and emtricitabine combination
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in care, at high risk of HIV infection: Patients in care, at high risk of HIV infection, according to the criteria defined by the French Ministry Of Health for the use of FTC / TDF in PreP (men who have sex with men, transgender, heterosexual women migrants or not, sex workers (sexual intercourse in exchange for money, drugs, housing, food), intravenous drug users) HIV-negative, exposed by their sexual practices to a high risk of HIV infection.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire should be completed by the patient the day of inclusion. Health data will be collected in patients medical file from inclusion to the date of the end of study (i.e. no follow-up for the last patient included and a maximum of three years of follow-up for the first patient included).

SUMMARY:
Despite the implementation of a national strategy to prevent the transmission of the human immunodeficiency virus (HIV) combining prevention campaigns, condom use, early detection of HIV infections and recommendations for treatment as soon as possible, the number of new HIV-infected patients per year in France does not decrease.

New HIV prevention strategies are therefore clearly needed. Since 2009, several studies have shown that tenofovir disoproxil fumarate and emtricitabine (TDF/FTC), an antiretroviral therapy combining two nucleoside reverse transcriptase inhibitors used for the treatment of patients seropositive for HIV, has preventive activity on HIV transmission. These results enabled the TDF/FTC to obtain in France an extension of the marketing authorization in March 2017 for preexposure prophylaxis (PrEP) of HIV transmission among patients at high risk of contamination.

Since the approval, many studies around the world investigate the use of PrEP in routine practice, highlighting its effectiveness in real life. These studies describe the population of patients who benefit from PrEP in order to adapt their multidisciplinary care but also track the transmission of other sexually transmitted infections to prevent their emergence, given the observed decline in condom use. However, these studies are limited to big cities while PrEP is accessible in all territories.

The Rhône-Alpes region is one of the three French regions that has been the most involved in the implementation of PrEP, one year after the FTC/TDF approval in France. Given the geographical position of the investigators, both in province and close to Switzerland, where the FTC/TDF is not authorized for PrEP, and the non-university nature of five of the six involved hospitals, the investigators would like to determine the profile of patients consulting in this region to benefit from PrEP. This analysis will also determine if the population at risk of the "Alpine Arc" region is similar to that observed in the other cohorts in order to adapt patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patient having initiated or wishing to initiate PrEP according to the recommendations of the French High Authority of Health in the centers involved in the collection of data
* Patient informed of the study and having indicated his non opposition for the collection of his health data

Exclusion Criteria:

* Wardship patient
* Patient under curatorship
* Patient unable to give his non-opposition to the use of his health data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in care, at high risk of HIV infection, according to the criteria defined by the French Ministery Of Health for the use of FTC / TDF in PreP (men who have sex with men, transgender, heterosexual women migrants or not, sex workers (sexual intercourse in exchange for money, drugs, housing, food), intravenous drug users) HIV-negative, exposed by their sexual practices to a high risk of HIV infection.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Questionnaire | one day
  Characterisation of people asking for HIV prophylaxis (either implementation or follow-up) : age, gender, past medical history and risk-taking of patients consulting for PrEP

SECONDARY OUTCOMES:
Incidence of HIV infections in PrEP patients and their management | up to 3 years
  Incidence of HIV infection in different key populations starting PrEP and according to PrEP use pattern (continuous or on demand) Frequency of HIV resistance to antiretrovirals (especially FTC and tenofovir - mutations at positions 184, 65, and 70 on the reverse transcriptase gene) Evaluation of the date of contamination (primary infection)
Use of post-exposure treatment | up to 3 years
  Frequency of use of post-exposure treatment, reasons, tolerance and effectiveness
Adherence to PrEP | one month
  Number of tablet consumption in the last month before the visit to the hospital as reported by the patients during the visit according to PrEP use pattern (continuous or on demand)
Tolerance of PrEP | up to 3 years
  Number of Clinical and Biological Adverse Events Considered Related to PrEP and Serious (CTCAE v5.0, grade 3 and 4), or Those Leading to Discontinuation of PrEP
Impact of PrEP on the evolution of risky sexual behavior | 4 weeks
  Number of sexual partners in the 4 weeks prior to visits Analysis of the last sex before the visit (type of sexual intercourse, use of the condom and / or PrEP)
Sexually Transmitted Infections | up to 3 years
  Number of Sexually Transmitted Infections (syphilis, chlamydia, gonococci, hepatitis C) acquired under PrEP and evolution during follow-up
Impact of PrEP in HIV and hepatitis screening | one day
  Number of patients for HIV and/or Hepatitis positive at first consultation

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Janssen, MD, Principal Investigator — CH Annecy Genevois
Locations (6):
- France (6):
  - CH de Belley, Belley
  - CH Métropole Savoie, Chambéry
  - CH Alpes Léman, Contamine-sur-Arve
  - CHU Grenoble, La Tronche
  - Centre Hospitalier Annecy Genevois, Metz-Tessy
  - CH de Sallanches, Sallanches

IPD SHARING:
Plan to Share IPD: Undecided